CLINICAL TRIAL: NCT02999399
Title: Assessing the Effect of Glucobrassicin-Rich Brussels Sprouts on the Metabolism of Deuterated Phenanthrene: Developing Food-Based Chemoprevention of Tobacco-Related Lung Cancer
Brief Title: Glucobrassicin-Brussel Sprout Effect on D10 Phe Metabolism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1610M96281
Record Dates: First submitted 2016-11-15; First posted 2016-12-21 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Smoking
Keywords: Smoker; Former smoker
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [D10]phe and Brussels sprouts (Experimental): All subjects are given 1 microgram [D10]phe before and after consuming Brussels sprouts once daily for 7 consecutive days.
  Interventions: Other: Brussel Sprouts; Drug: Deuterated Phenanthrene

INTERVENTIONS:
Other: Brussel Sprouts — Subjects are given ~150 g of Brussels sprouts once daily for 7 consecutive days.
Drug: Deuterated Phenanthrene — Subjects are given 1 microgram of deuterated phenanthrene [D10]phe at baseline and after 7 days of Brussels sprout consumption. Urine is collected for 6 hours after each dose.

SUMMARY:
To determine whether glucobrassicin-rich Brussels sprouts can favorably modify the metabolism of the polycyclic aromatic hydrocarbon deuterated phenanthrene ([D10]phe) in current and former smokers

DETAILED DESCRIPTION:
Subjects will be given 1 microgram of [D10]phe, and all urine will be collected for 6 h afterwards to quantify baseline levels of [D10]phenanthrene tetraol ([D10]pheT) and [D10]phenanthrols ([D10]HOP). Within 3 days of this baseline measurement, subjects will consume 200 micromoles of glucobrassicin in the form of raw Brussels sprouts (~200-300 grams) at the study center once daily for 7 consecutive days. Urine will be collected for 24 h after vegetable consumption on days 3 ± 1 and 6 of the feeding intervention for 3,3'-diindolylmethane (DIM) quantification. On day 7 of the feeding intervention, a second dose of 1 microgram of [D10]phe will be administered at the study center after vegetable consumption, followed by another 6 h urine collection.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years old
* Current or former smoker by self-report
* Willing to abstain from cruciferous vegetable consumption other than the study vegetable during the study period
* Able to understand the experimental nature of the study and provide informed consent
* Negative urine pregnancy test for women of childbearing potential within 7 days of baseline [D10]phe dosing

Exclusion Criteria:

* Chronic proton pump inhibitor, H2-blocker (i.e., ranitidine, famotidine), and/or calcium carbonate use
* History of gastric bypass surgery, gastric banding, bowel resection, malabsorption syndromes such as celiac sprue or pancreatic insufficiency, or other conditions that may affect gastric absorption
* Current use of tobacco products other than cigarettes (i.e. snuff, snuz, smokeless tobacco, cigars, pipes) or use of these products within 3 months of study registration
* Major or chronic medical disease, including heart disease, poorly controlled diabetes, etc., to be adjudicated by the principal investigator
* Women who are pregnant, intend to become pregnant within 3 months of the study period, or who are breastfeeding
* Current or recent (within 12 months) problems with drug use or alcohol dependence by self-report Antibiotic use within 2 months of study enrollment or during the study by self-report Alcohol dependence, abuse, or history of dependence/abuse by self-report Vegetarians
* History of respiratory tract cancer
* Use of metronidazole or antabuse during the study
* Taking ibuprofen, naproxen, other NSAIDs, steroids (except inhaled steroids) within 14 days of study registration
* Allergy to Brussels sprouts

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Change in [D10]phenanthrene tetraol | 7 days
  Compare level of urinary [D10]phenanthrene tetraol before and after 7 days of Brussels sprout consumption.

SECONDARY OUTCOMES:
Change in [D10]phenanthrols | 7 days
  Compare level of urinary [D10]phenanthrene phenanthrols before and after 7 days of Brussels sprout consumption.
Change in [D10]phenanthrene tetraol:[D10]phenanthrol ratio | 7 days
  Compare level of urinary [D10]phenanthrene phenanthrols before and after 7 days of Brussels sprout consumption.

OTHER OUTCOMES:
Urinary 3,3'-diindolylmethane (DIM) | Day 3 and Day 6
  Urinary DIM will be quantified after Brussels sprout consumption on day 3 and day 6 of the feeding intervention for urinary DIM quantification

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Fujioka, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States